CLINICAL TRIAL: NCT02439645
Title: A Registry to Determine the Clinical and Genetic Risk Factors for Torsade De Pointes
Acronym: BA-TdP
Status: Terminated | Type: Observational
Why Stopped: Study was terminated lack of recruitment, small number of eligible cases (11 enrolled, 1 found ineligible after enrollment), unlikely to be able to achieve study goals due to low recruitment.
Sponsor: Massachusetts General Hospital (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency); Beth Israel Deaconess Medical Center (Other); Brigham and Women's Hospital (Other); Boston University (Other); Mayo Clinic (Other); The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Christopher Newton-Cheh, MD, Overall Principal Investigator, Massachusetts General Hospital
Other Study IDs: 2013P001531
Record Dates: First submitted 2015-05-05; First posted 2015-05-12 (Estimated); Last update posted 2021-12-03 (Actual); Status verified 2021-11

CONDITIONS: Long qt Syndrome; Torsade de Pointes
Keywords: genetic research
MeSH Terms: conditions — Long QT Syndrome; Torsades de Pointes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Biospecimen Retention: Samples With DNA — Blood samples from patients with a history of torsade de pointes.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is a registry to examine genetic and clinical predictors of torsade de pointes events.

DETAILED DESCRIPTION:
BACKGROUND AND SIGNIFICANCE Drug-induced long QT syndrome (LQTS), and the subsequent fatal arrhythmia torsade de pointes (TdP), is an important side effect associated with the use of a number of medications. Prolongation of the QT interval is the most common cause of withdrawal of medications already on the market, and despite the relatively rarity with non-cardiovascular drugs, the public health impact is magnified by the fact that drug-induced TdP can occur with medications used for benign conditions, such as allergic rhinitis. The QT interval is heritable, and a number of common genetic variants have been associated with QT interval in large population studies.

Although common genetic variants associated with sudden cardiac death have been identified, studies specifically identifying variants associated with drug-induced LQTS and TdP are limited. Smaller studies have suggested that variants of genes associated with QT interval duration in the population in general are also associated with the risk of drug-induced QT prolongation and TdP, but larger studies are needed. Moreover, an improved ability to predict the causes of TdP requires a careful search for clinical factors associated with TdP compared to controls.

RESEARCH DESIGN AND METHODS

A. Study Design and Enrollment: We propose to conduct a multi-center research study to examine known and explore potentially unknown genetic and clinical predictors of torsade de pointes (TdP) also known as acquired long QT syndrome (LQTS) through creation of a registry. Any patient with a documented history of a torsade de pointes (TdP) event will be eligible. Patients must be able to understand the risks of genetic testing, and be willing to undergo a venipuncture for blood collection for genotyping. Exclusion criteria include inability to provide informed consent. We plan to enroll a total of 200 study participants total across all participating centers. Massachusetts General Hospital will be the coordinating center of this multi-center study of medical institutions within the greater Boston and New England area. In a substudy to take place at MGH, subjects will be invited to have a punch biopsy of the skin to allow creation of inducible pluripotent stem cells that can be differentiated into cardiomyocytes for further characterization of the repolarization phenotype.

B. Study Procedures: We will screen patients for enrollment including both retrospective (event prior to the start of the study) and prospective (event following the start of the study) components. Patients will be identified by investigators based on clinical characteristics, and following explanation of the study by co-investigators, will be asked about participation either during routine scheduled follow-up (for retrospective cases) or at the sentinel event. Investigators will complete a data collection form for each patient, which will include contact information, demographic information, clinical information, family history and pedigree, and all electrocardiography information available (12-lead ECGs, rhythm strips and summary reports). No information about mental illness will be collected. Patients will then undergo venipuncture, and four 5mL blood samples will be collected for genotyping and plasma analysis. For patients who are willing, a 3mm punch biopsy from the shoulder, upper thigh, small of the back, or buttock (subject's choice) will be obtained for fibroblast culture. Patients who are recruited at non-MGH sites will have a visit to MGH scheduled in order to obtain the skin biopsy. Induced pluripotent stem cells will be made from the fibroblast cultures and differentiated to cardiomyocytes in order to assess the cellular phenotype. Patients will also be consented for future re-contact about additional data, information, or samples needed for analysis. All clinical information and samples (including DNA and blood) collected at participating centers will be transferred to Dr. Newton-Cheh at MGH for storage and analysis.

ELIGIBILITY:
For simplicity, we will plan to include all possible cases of TdP meeting criteria (see below) into the registry.

Exclusion criteria include:

1. age <18 years old
2. inability to obtain informed consent from the patient or a family member
3. no exclusion on the basis of race or gender.

Inclusion criteria include:

torsade de pointes clinical syndrome according to one of the following three clinical criteria:

1. Definite TdP: At least 3 beats of polymorphic ventricular tachycardia (VT) or ventricular fibrillation (VF) on a 12-lead ECG or rhythm strip with documented QTc > 450 ms in men or QTc > 470 in women (excluding patients with conduction block or AF at baseline, see below) prior to arrhythmic event.
2. Probable TdP: At least 3 beats of polymorphic VT or VF on a 12-lead ECG or rhythm strip with QTc > 450ms (men) or 470ms (women) after the event, or polymorphic VT or VF episode not meeting criteria for 'definite TdP' but determined by the adjudicating physician to be likely TdP. For patients having a cardiac arrest, at least 1 hour after restoration of normal rhythm or after secondary hypoxia or electrolyte abnormalities have been ruled out (confounders of QT prolongation often seen post-arrest47) will be required.
3. Possible TdP: Unexplained syncope in a patient presenting with QTc > 450ms (men) or 470ms (women).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient in which informed consent can be obtained, with a history of torsade de points (see below designation).
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2013-10; Primary Completion 2019-07-26 (Actual); Study Completion 2019-07-26 (Actual)

PRIMARY OUTCOMES:
Torsade de pointes arrhythmia events | Participants will be followed for the time to obtain consent, clinical information and biospecimens (typically < 1 day)
  1. Definite TdP: At least 3 beats of polymorphic ventricular tachycardia (VT) or ventricular fibrillation (VF) on a 12-lead ECG or rhythm strip with documented QTc > 450 ms in men or QTc > 470 in women (excluding patients with conduction block or AF at baseline, see below) prior to arrhythmic event.
  2. Probable TdP: At least 3 beats of polymorphic VT or VF on a 12-lead ECG or rhythm strip with QTc > 450ms (men) or 470ms (women) after the event, or polymorphic VT or VF episode not meeting criteria for 'definite TdP' but determined by the adjudicating physician to be likely TdP. For patients having a cardiac arrest, at least 1 hour after restoration of normal rhythm or after secondary hypoxia or electrolyte abnormalities have been ruled out (confounders of QT prolongation often seen post-arrest47) will be required.
  3. Possible TdP: Unexplained syncope in a patient presenting with QTc > 450ms (men) or 470ms (women).

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Newton-Cheh, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (4):
- United States (4):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston University Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - West Roxbury VA Medical Center, West Roxbury, Massachusetts